CLINICAL TRIAL: NCT01641055
Title: A 8 wk Study to Compare the Effects of Proteins Various Fish Species (Salmon, Herring, Cod) and Milk on Glucose Regulation in Overweight and Obese Adults.
Brief Title: A Study of the Effects of Fish Protein Intake on Glucose Regulation in Overweight and Obese Adults.
Acronym: FISK3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: BlueProtein (Unknown); NutriMar (Unknown)
Responsible Party: Principal Investigator, Oddrun Anita Gudbrandsen, PhD, University of Bergen
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2011/572
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Allergen M protein, codfish; Milk Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Salmon protein hydrolysate (Experimental)
  Interventions: Dietary Supplement: Salmon protein hydrolysate
- Herring protein hydrolysate (Experimental)
  Interventions: Dietary Supplement: Herring protein hydrolysate
- Cod protein (Sham Comparator)
  Interventions: Dietary Supplement: Cod protein
- Milk protein (Placebo Comparator)
  Interventions: Dietary Supplement: Milk protein

INTERVENTIONS:
Dietary Supplement: Salmon protein hydrolysate — 2.5g salmon protein hydrolysate per day for 8wk.
  Arms: Salmon protein hydrolysate
Dietary Supplement: Herring protein hydrolysate — 2.5g herring protein hydrolysate per day for 8wk.
  Arms: Herring protein hydrolysate
Dietary Supplement: Cod protein — 2.5g cod protein per day for 8wk.
  Arms: Cod protein
Dietary Supplement: Milk protein — 2.5g milk protein per day for 8wk.
  Arms: Milk protein

SUMMARY:
The purpose of this study is to compare the possible health benefits of intake of proteins from salmon, herring, cod and milk on glucose tolerance in overweight and obese adults. Overweight and obese subjects often have reduced glucose tolerance, and previous findings from a study on cod proteins suggested that glucose tolerance was improved.

DETAILED DESCRIPTION:
Participants receive 2.5g protein per day for 8 weeks as tablets.

ELIGIBILITY:
Inclusion Criteria:

* BMI above 27 kg/m2
* healthy

Exclusion Criteria:

* fasting blood glucose above 7 mM
* medication that affects blood glucose, lipids and inflammatory status
* pregnancy or breastfeeding
* allergies to fish or milk
* intentional weight loss and large fluctuation in body weight
* a high consumption of fish
* an extreme diet
* use of fish oil, n-3 or multivitamin supplements

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Glucose regulation | 8 weeks
  Glucose will be measured in fasting and postprandial samples

SECONDARY OUTCOMES:
Changes in serum insulin, insulin C-peptide, non-esterified fatty acids, lipids, adiponectin, leptin and fatty acid composition | 8 weeks
Changes in serum and urine concentrations of amino acids and their metabolites | 8 weeks
Changes in serum concentrations of vitamins | 8 weeks
Comparisons of metabolites and co-factors involved in one-carbon metabolism in serum and urine | 8 weeks
  Concentrations of relevant metabolites and co-factors were measured in serum and urine

CONTACTS AND LOCATIONS:
Overall Officials: Oddrun A Gudbrandsen, PhD, Principal Investigator — University of Bergen
Locations (1):
- Institute of Medicine, University of Bergen, Bergen, Norway

REFERENCES:
- [Derived] Hovland IH, Leikanger IS, Stokkeland O, Waage KH, Mjos SA, Brokstad KA, McCann A, Ueland PM, Slizyte R, Carvajal A, Mellgren G, Remman T, Hogoy I, Gudbrandsen OA. Effects of low doses of fish and milk proteins on glucose regulation and markers of insulin sensitivity in overweight adults: a randomised, double blind study. Eur J Nutr. 2020 Apr;59(3):1013-1029. doi: 10.1007/s00394-019-01963-0. Epub 2019 Apr 10. PMID 30972484